CLINICAL TRIAL: NCT00327704
Title: Multicenter, Prospective, Randomized, Controlled Open Study Albumin 20% Versus Saline
Brief Title: Early Albumin Resuscitation During Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Jean-Paul MIRA, Professor, Cochin Hospital, Paris France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFB N°ALBU-0503
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Septic Shock
Keywords: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Albumins; Sodium Chloride

ARMS (2):
- Albumin (Active Comparator)
  Interventions: Drug: albumin
- Saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: albumin — albumin 20% 100 ml/8 hours for 3 days
  Other Names: Vialebex
  Arms: Albumin
Drug: saline — saline 100 ml/8hours for 3 days
  Arms: Saline

SUMMARY:
Objective: To determine whether the early administration of albumin as an expander and antioxidant would improve survival on the 28th day for septic shock patients.

Design: Prospective, multicenter, randomized, controlled versus saline, stratified on nosocomial infection and center.

Setting: 27 Intensive Care Units (ICU) in France

Coordinator: Pr J.P. Mira and Dr J. Charpentier - Cochin Hospital- Paris

Patients: 800 patients could be included during the first 6 hours of their septic shock.

DETAILED DESCRIPTION:
The primary outcome: Mortality during the 28 day period after randomization. The secondary outcomes: Evaluation of SOFA score, ventilator-free days, dialysis free days, catecholamine free days, days of hospitalisation, incidence of nosocomial infections.

The albuminemia of all patients is requested before the treatment until Day 4 post treatment.

The treatment is: Vialebex 20% 100ml every 8 hours during 3 days versus saline 100ml every 8 hours during 3 days.

The first patient will be in July 2006, the last patient expected is on July 2009.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Septic shock < 6 hours
* Agreement of patients

Exclusion Criteria:

* Allergy to albumin
* Weight > 120 kg
* Non septic shock
* Burned
* Cirrhosis
* Albumin perfusion 48 hours before randomization
* Pregnant women
* Cardiac dysfunction New York Heart Association (NYHA) 3 or 4
* Patients with therapeutic limitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Mortality, any cause, during the 28 day period after randomization | day 28

SECONDARY OUTCOMES:
Evaluation of sequential organ failure assessment (SOFA) score | ICU period
catecholamine free days | day 28
incidence of nosocomial infection | ICU period
mortality at 90 days | day 90
length of ICU hospitalisation | ICU discharge
length of total hospitalisation | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jean P Mira, Professor, Study Chair — Cochin Hospital; Julien Charpentier, Doctor, Study Director — Hôpital Cochin
Locations (1):
- Cochin Hospital, Paris, Paris, France